CLINICAL TRIAL: NCT05265702
Title: Effectiveness of Non-Invasive Neuromodulation in Children With Neurodevelopmental Disorders to Improve Constipation and Sleep Quality
Brief Title: Non-Invasive Neuromodulation in Children With Neurodevelopmental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Principal Investigator, University of Las Palmas de Gran Canaria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NESA SJD
Record Dates: First submitted 2022-02-18; First posted 2022-03-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Neurodevelopmental Disorders
Keywords: physical therapy modality; Electric Stimulation Therapy; Child Development Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders; Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-invasive Neuromodulation (Experimental): Non-invasive Neuromodulation Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7 level.
  Interventions: Device: Non-invasive Neuromodulation

INTERVENTIONS:
Device: Non-invasive Neuromodulation — The electrodes will be placed with the help of gloves and adapted socks for 1 hour, twice a week, until 12 intervention sessions are completed. In addition, depending on the session, an adhesive electrode will be placed at the level of C7. Characteristics of microcurrents: pulsed monophasic rectangular wave with a pulse of 1.3 s and pause of 300 ms, voltage 3 millivolt and intensity 0.5 μA.

SUMMARY:
Children with neurodevelopmental disorders have a delay in acquiring the skills that are assumed considering the phases of typical psychomotor development. Added to this difficulty and main element of concern on the part of their families, there are another series of signs that appear with some frequency and that, despite being unnoticed against other major problems represent basic and fundamental factors in the correct development and performance such as constipation problems and sleep disorders.

The aim of the study consists of to evaluate the effectiveness and safety of the non-invasive neuromodulation device applied in people with neurodevelopmental disorders, in relation to constipation problems and in the quality of sleep.

DETAILED DESCRIPTION:
While the application is being sent to the ethics committee, we will hold a series of informative talks for the centre's staff who, in one way or another, will be involved in the development of the project.

At the same time, information letters will be sent to the parents or legal representatives of the children who will a priori be part of the project, as well as the corresponding informed consent. In addition, they will be sent the screening documents that will allow us to confirm if the selected subject has constipation problems and/or sleep disorders.

The intervention period per subject will be 12 sessions, distributed in three sessions per week (Monday, Wednesday, and Friday), estimating that the intervention can be completed after one month.

During school hours, the participants will receive their own treatment, agreed by their multidisciplinary team with common and personal objectives for the subjects, so that there will be no interruption of their usual routine.

Two weeks after the intervention, a new assessment will be carried out to assess whether the possible changes recorded during the intervention phase have been maintained.

ELIGIBILITY:
Inclusion Criteria:

* Sensory-motor alteration.
* Be schooled in the Center of the City San Juan de Dios of Las Palmas de Gran Canaria.
* Meet the criteria established by the Rome IV constipation scale.
* Informed consent signed by the family, guardian or legal representative.

Exclusion Criteria:

* No contraindications to treatment with NXSignal: Pacemaker, internal bleeding, do not apply electrodes on skin in poor condition, with ulcerations or wounds, acute febrile processes, acute thrombophlebitis and/or phobia to electricity.
* Epilepsia.
* Subjects who modify eating habits and/or water intake.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Change in stool characteristics from baseline at a month and a half | Baseline and up to 1 month, and two weeks after intervention
  A daily evaluation will be carried out both number of stools, as well as the type of stools following the criteria established by the Bristol Stool Form Scale. It is widely used as a research tool to assess the efficacy of treatments for various diseases of the intestine. The chart is used to describe the shapes and types of stool. It is also used as a tool to diagnose constipation, diarrhea, and irritable bowel syndrome.
  It is a medical aid designed to classify faeces into seven groups: Types 1 and 2 indicate constipation, types 3 and 4 are considered healthy stool, while types 5 to 7 suggest diarrhea and urgency.
  Each person will have different bowel habits, but the important thing is that your stools are soft and easy to pass, like types 3 and 4.
Change in sleep diary from baseline at a month and a half | Baseline and up to 1 month, and two weeks after intervention
  The sleep diary is easy to complete and gives us a global vision of sleep for several days. It facilitates the calculation of hours of sleep and nocturnal awakenings.
  The person who registers indicates the number of hours of sleep

SECONDARY OUTCOMES:
Frequency of defecation from baseline at a month and a half | Baseline and up to 1 month, and two weeks after intervention
  It will be recorded in number of times in which the participant defecates.

CONTACTS AND LOCATIONS:
Overall Officials: Aníbal Báez-Suárez, PhD, Principal Investigator — University of Las Palmas de Gran Canaria
Locations (1):
- Aníbal Báez Suárez, Las Palmas de Gran Canaria, Palmas, Las, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thapar A, Cooper M, Rutter M. Neurodevelopmental disorders. Lancet Psychiatry. 2017 Apr;4(4):339-346. doi: 10.1016/S2215-0366(16)30376-5. Epub 2016 Dec 13. PMID 27979720
- [Result] Ambartsumyan L, Rodriguez L. Gastrointestinal motility disorders in children. Gastroenterol Hepatol (N Y). 2014 Jan;10(1):16-26. PMID 24799835
- [Result] Sood R, Ford AC. Diagnosis: Rome IV criteria for FGIDs - an improvement or more of the same? Nat Rev Gastroenterol Hepatol. 2016 Sep;13(9):501-2. doi: 10.1038/nrgastro.2016.110. Epub 2016 Jul 13. No abstract available. PMID 27407043
- [Result] Robertson J, Baines S, Emerson E, Hatton C. Constipation management in people with intellectual disability: A systematic review. J Appl Res Intellect Disabil. 2018 Sep;31(5):709-724. doi: 10.1111/jar.12426. Epub 2017 Nov 23. PMID 29168259
- [Derived] Baez-Suarez A, Padron-Rodriguez I, Castellano-Moreno E, Gonzalez-Gonzalez E, Quintana-Montesdeoca MP, Medina-Ramirez RI. Application of non-invasive neuromodulation in children with neurodevelopmental disorders to improve their sleep quality and constipation. BMC Pediatr. 2023 Sep 15;23(1):465. doi: 10.1186/s12887-023-04307-4. PMID 37715152